CLINICAL TRIAL: NCT02622984
Title: Remote Brief Intervention and Referrals to Treatment Service for Alcohol
Acronym: RBIRT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Polaris Health Directions (Industry)
Collaborators: University of Massachusetts, Worcester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2R42AA02203503
Record Dates: First submitted 2015-11-19; First posted 2015-12-07 (Estimated); Last update posted 2021-03-10 (Actual); Status verified 2020-03

CONDITIONS: Alcohol Abuse, Alcohol Dependence
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RBIRT (Experimental): Telehealth model or the remote administration of SBIRT, a short term, brief intervention and referral to treatment for alcohol abuse.
  Interventions: Behavioral: RBIRT
- SBIRT (Active Comparator): Face-to-face intervention and referral to treatment for alcohol abuse.
  Interventions: Behavioral: SBIRT

INTERVENTIONS:
Behavioral: RBIRT — Intervention group will receive the telehealth or remote behavior intervention and referral for substance use (RBIRT). Other group will receive treatment as usual which is SBIRT.
  Arms: RBIRT
Behavioral: SBIRT — Face to face standard intervention considered "treatment as usual."
  Arms: SBIRT

SUMMARY:
The traditional paradigm that relies upon training physicians and nurses or uses on-site interventionists to perform screening, brief intervention, and referral to treatment (SBIRT) for alcohol has proven unsustainable in most clinical settings. The Remote Brief Intervention and Referral to Treatment (R-BIRT) for alcohol is an innovative telehealth service model with potential to improve public health through evidence based counseling for patients who exceed the NIAAA low risk drinking limits or have evidence of an Alcohol Use Disorder with professional and self-help treatment. For those that are appropriate, the R-BIRT service will provide facilitated referrals to specialized alcohol abuse treatment. The service model is being studied in the emergency department (ED) setting to demonstrate its utility in a medical setting with a very high prevalence of risky alcohol use and Alcohol Use Disorders; however, the model is relevant and will be accessible to a broad array of healthcare settings, including primary care practices. Our new model, the R-BIRT, challenges the prevailing paradigm and offers the promise of not only clinical efficacy but increased cost effectiveness as well.

DETAILED DESCRIPTION:
Significance: The USPHSTF, SAMHSA, CDC, and NIAAA have affirmed the importance of screening in medical settings for alcohol consumption that exceeds the NIAAA low risk limits, brief educational and motivational counseling for those who screen positive or have other evidence of an Alcohol Use Disorder, and, when appropriate, referral to treatment (SBIRT). However, translation to clinical practice continues to be elusive. Polaris Health Directions (Small Business) and the University of Massachusetts Medical School (Research Institute) have partnered to solve this problem by creating the Remote Brief Intervention and Referral to Treatment service for alcohol (R-BIRT), a telehealth service for delivering evidence based alcohol brief interventions and referral to treatment during a medical encounter in a cost-effective, sustainable way.

Investigators: The investigators have extensive expertise in SBIRT for alcohol (Boudreaux, Bernstein); telehealth (Boudreaux); development, testing, and marketing of behavioral intervention technologies (Boudreaux, Harralson); comparative effectiveness trial design and analysis (Barton); and health economics (Sachs). Combined, the team has over 100 publications related to SBIRT and constituent technology domains.

Innovation: This Phase 2 STTR will pioneer telehealth delivery of SBIRT for alcohol. It will be flexible enough for a variety of medical settings, and will develop and expand software capable of facilitating both telehealth and in-person SBIRT delivery models. It will further innovate SBIRT research and clinical practice by exploring mechanisms of action, an objective rarely incorporated into SBIRT studies.

Approach: The design is a two arm, single blind (outcomes assessor), randomized, non-inferiority trial. Emergency department (ED) patients (n=356) who drink above the NIAAA low risk limits or have evidence of an Alcohol Use Disorder will be randomized to the telehealth model (R-BIRT) or a gold-standard in-person intervention (SBIRT) and followed for 6 months post-visit using a multi-method outcomes attainment plan. The study will establish the non-inferiority of the telehealth model compared to the in-person model in reducing alcohol use and alcohol related consequences, while showing that the telehealth model is the more cost effective of the two. Mechanisms of action, including patient knowledge of low risk drinking limits, motivation, self-efficacy, substance abuse treatment initiation, and self-help program engagement, will be examined.

Environment: With the success of the R-BIRT Phase 1 and other relevant projects, including previous large scale Phase 2 STTR clinical trials, Polaris and UMass have clearly established their capability of successfully carrying out this study, disseminating its results, and marketing the final product.

Impact: Because alcohol misuse, abuse, and dependence carries an enormous burden in both human suffering and healthcare costs, a strategy that provides high quality, evidence based care in a manner that is more cost effective and easier than existing models has potential to exert a substantial impact on public health.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older.
* Presenting for care to the UMass Emergency Department.
* Screens positive for alcohol use above the NIAAA age and gender matched low risk drinking limits.
* AUDIT-10 score greater than 8 suggesting risk for an Alcohol Use Disorder.

Exclusion Criteria:

* Altered mental status (not alert, not oriented, psychotic, persistent intoxication).
* Patients who present as initially intoxicated but who are no longer intoxicated later in the visit can be approached.
* Currently in alcohol treatment.
* DAST-10 score greater than 3.
* Currently in state custody or pending legal action that might lead to imprisonment.
* Cannot paraphrase the study requirements.
* No reliable telephone access.
* Does not speak English.
* Already enrolled into the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Change in alcohol use across the study period compared to baseline. | 1,3, 6 months post Emergency Department (ED) visit
  Consistent with the latest standards in ED SBIRT research, alcohol use will be measured by a one-week Timeline Follow-back (TLFB), which is a validated procedure wherein participants report the number of drinks they consumed each day for the past seven days using a protocol that facilitates recall. This will allow computation of drinks/week and drinking above the NIAAA low risk drinking limits.

SECONDARY OUTCOMES:
Changes in alcohol related consequences across the study period compared to baseline. | 1,3,6 months post ED visit
  Alcohol-related consequences will be measured by the Short Inventory of Problems (SIPs+6).
Changes in acute healthcare utilization at 6 months compared to baseline. | 6 months post ED visit
  The Cornell Services Index will be used to ascertain all outpatient and inpatient healthcare use, including substance abuse treatment. It will be modified to also assess self-help program engagement, such as Alcoholics Anonymous. Per our standard procedures used in other studies, self-reported substance abuse treatment initiation will be validated by contacting the treating provider.
Compare the costs of both interventions: SBIRT and RBIRT. | 6 months post ED visit
  Intervention Cost data will be estimated by standard costing methods taking into account all of the costs associated with delivery of both interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Edwin D Boudreaux, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States